CLINICAL TRIAL: NCT01208831
Title: An East Asian Phase I, Multicenter, Open-label, Dose-escalation Study of Oral LDE225 in Patients With Advanced Solid Tumors
Brief Title: An East Asian Study of LDE225
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDE225X1101
Record Dates: First submitted 2010-09-21; First posted 2010-09-24 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2016-04

CONDITIONS: Advanced Solid Tumor Cancers; Medulloblastoma; Basal Cell Carcinoma
Keywords: Advanced tumors; hedgehog; smoothened inhibitor
MeSH Terms: conditions — Medulloblastoma; Carcinoma, Basal Cell | interventions — sonidegib

ARMS (1):
- LDE225 (Experimental)
  Interventions: Drug: LDE225

INTERVENTIONS:
Drug: LDE225

SUMMARY:
The purpose of this study is to determine Maximum Tolerated Dose (MTD) or recommended phase II dose of LDE225 when administered orally to two adult patient groups of East Asian (i.e., Japanese and Chinese/Taiwanese) with advanced solid tumors that have progressed despite standard therapy or for which no standard therapy exists.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of advanced solid tumor (including medulloblastoma and basal cell carcinoma)
* blood work criteria

Exclusion Criteria:

* patients with history of brain tumor (except recurrent medulloblastoma) or brain metastases
* positive HIV, hepatitis B or C
* impaired intestinal function
* impaired heart function
* pregnant or breast-feeding women

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
determine maximum tolerated dose of single agent LDE225 | 28 day cycles

SECONDARY OUTCOMES:
characterize safety and tolerability | 28 day cycles
characterize pharmacokinetics (PK) of single and repeated doses of LDE225 | 28 day cycles
assess preliminary anti-tumor activity | 28 day cycles

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Novartis Investigative Site, Hong Kong, Hong Kong
- Japan (2):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kobe, Hyōgo
- Novartis Investigative Site, Taipei, Taiwan

REFERENCES:
- [Derived] Minami H, Ando Y, Ma BB, Hsiang Lee J, Momota H, Fujiwara Y, Li L, Fukino K, Ito K, Tajima T, Mori A, Lin CC. Phase I, multicenter, open-label, dose-escalation study of sonidegib in Asian patients with advanced solid tumors. Cancer Sci. 2016 Oct;107(10):1477-1483. doi: 10.1111/cas.13022. Epub 2016 Sep 24. PMID 27467121
- See also: Results for CLDE225X1101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=12324